CLINICAL TRIAL: NCT06566950
Title: Effectiveness of Blood Flow Restriction Training on Muscle Morphology and Prevention of Patellofemoral Pain Syndrome and Anterior Cruciate Ligament Injury
Brief Title: BFR Training on Muscle Morphology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, I Putu Gde Surya Adhitya, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1791/UN14.2.2.VII.14/LT.2024
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Blood Flow Restriction Training; Eccentric Training; Muscle Morphology; Patellofemoral Pain Syndrome; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low load-BFRt (Experimental): 70% of the arterial occlusion pressure and 30% of the maximum repetition rate
  Interventions: Procedure: Low load-BFRt
- Sham Low load-BFRt (Sham Comparator): 10% of the arterial occlusion pressure and 30% of the maximum repetition rate
  Interventions: Procedure: Sham Low load-BFRt
- High load-Eccentric training (Active Comparator): 70% of the maximum repetition rate
  Interventions: Procedure: High load-Eccentric training

INTERVENTIONS:
Procedure: Low load-BFRt — The participants' two legs will be subjected to 70% arterial occlusion pressure when the physical therapist applies the BFR cuffs. After that, participants will be required to complete eccentric exercises with a maximum repetition count of 30%, such as stairs, single leg squat, and single leg deadlift.
  Arms: Low load-BFRt
Procedure: Sham Low load-BFRt — The participants' two legs will be subjected to 10% arterial occlusion pressure when the physical therapist applies the BFR cuffs. After that, participants will be required to complete eccentric exercises with a maximum repetition count of 30%, such as stairs, single leg squat, and single leg deadlift.
  Arms: Sham Low load-BFRt
Procedure: High load-Eccentric training — The physical therapist will instruct the participants to complete eccentric exercises at a maximum of 70% repetitions, such as stairs, single leg squat, and single leg deadlift.
  Arms: High load-Eccentric training

SUMMARY:
This randomized clinical trial study compares high-load eccentric training (HL-Et), sham LL-BFRt, and low-load blood flow restriction (LL-BFRt) in sportsmen. The primary inquiries it seeks to address are:

Is LL-BFR superior to HL-Et and sham LL-BFRt in terms of improving muscle morphology? Is LL-BFR a more effective Patellofemoral Pain Syndrome and ACL injury preventive than HL-Et and sham LL-BFRt?

The three intervention groups that will be randomly assigned to participants are LL-BFRt, sham LL-BFRt, and HL-Et. Participants are expected to carry out:

Participants in LL-BFRt will be required to perform LL eccentric training at 30% of their repetition maximum (RM) and 70% of their artery occlusion pressure (AOP). This training will include stairs, single leg squat, and single leg deadlift.

Participants in HL-Et will be required to perform LL eccentric training at 70% of their maximum number of repetitions (RM).

In order to determine whether muscular morphology and the prevention of Patellofemoral Pain Syndrome and ACL injury improve following the interventions and follow-up, researchers will compare LL-BFRt, sham LL-BFRt, and HL-Et.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 15 and 35
* Play level 1 sports (fight martial arts, basketball, futsal, and soccer) at least twice a week
* Never experienced an Patellofemoral Pain Syndrome or ACL injury before
* Never experienced a grade III sprain or strain
* Consent to participate in the study until its conclusion and provide informed consent.

Exclusion Criteria:

* Having a tumor, cancer, vena thromboembolic disease, obesity, diabetes, hypertension, anemia, and renal failure
* Disabilities or those who are disabled.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Muscle cross-sectional area | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the cross-sectional area of vastus medial obliques muscle and peroneus longus muscle.
Vastus medial obliques fiber angle | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the vastus medial obliques fiber angle.
Patella position | 8 weeks
  Using a musculoskeletal ultrasonography, researchers will determine the patella position.

SECONDARY OUTCOMES:
Incidence of patellofemoral pain syndrome | 1 year
  Researchers will determine the incidence of patellofemoral pain syndrome with the physical examination of grind test.
Incidence of anterior cruciate ligament injury | 1 year
  Researchers will determine the incidence of anterior cruciate ligament injury with the physical examination of Lachman's test.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical therapy laboratory, College of Medicine, Universitas Udayana and ROM Physiotherapy Private Clinic Denpasar, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No